CLINICAL TRIAL: NCT07397624
Title: Endoscopic Suture Gastroplasty (ESG) for Treatment of Obese Patients With Endometrial Cancer: a Prospective, Multicenter, Observational Study (ESG-ENDO)
Brief Title: Endoscopic Suture Gastroplasty (ESG) for Treatment of Obese Patients With Endometrial Cancer
Acronym: ESG-ENDO
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2025-016
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity increases the risk of endometrial cancer, with higher Body Mass Index (BMI) leading to a significant increase in both cancer risk and recurrence. Because of the excellent cancer-specific outcomes and preponderance of obesity-related complications, women with endometrial cancer are more likely to die of cardiovascular disease and other obesity-related illnesses than endometrial cancer itself. This makes an endometrial cancer diagnosis a critical moment to emphasizes the importance of actively managing the underlying issue of obesity in the endometrial cancer survivorship period.

Bariatric surgery has shown long-term benefits, including weight loss and reduction of obesity-related comorbidities, and has been linked to a decrease in endometrial cancer incidence. However, bariatric surgery has limitations, such as irreversibility and potential complications. Recent interest in less invasive methods, like bariatric endoscopy, shows promising results in achieving weight loss and improving metabolic profiles. Endoscopic procedures, such as Endomina Endoscopic suture gastroplasty (E-ESG), have shown effectiveness in weight loss and could offer a safer, more accessible alternative to surgery, in particular if associated to a lifestyle modifications program. Efficacy and safety of Bariatric endoscopy has been stressed within the recently published "Guideline of the Italian Society of Surgery of Obesity and Metabolic Diseases on Bariatric Endoscopy in the treatment of obesity and associated complications" that suggest the use of bariatric endoscopy in patients with class I obesity and in patients with class II obesity regardless of the presence of comorbidities, for the treatment of obesity.

This study aims to assess the feasibility and safety of the E-ESG procedure in treating obesity in women after curative treatment for endometrial cancer.

DETAILED DESCRIPTION:
Obesity increases the risk of endometrial cancer, with higher BMI leading to a significant increase in both cancer risk and recurrence. Because of the excellent cancer-specific outcomes and preponderance of obesity-related complications, women with endometrial cancer are more likely to die of cardiovascular disease and other obesity-related illnesses than endometrial cancer itself. This makes an endometrial cancer diagnosis a critical moment to emphasizes the importance of actively managing the underlying issue of obesity in the endometrial cancer survivorship period. Bariatric surgery has shown long-term benefits, including weight loss and reduction of obesity-related comorbidities, and has been linked to a decrease in endometrial cancer incidence. However, bariatric surgery has limitations, such as irreversibility and potential complications. Recent interest in less invasive methods, like bariatric endoscopy, shows promising results in achieving weight loss and improving metabolic profiles. Endoscopic procedures, such as Endomina Endoscopic suture gastroplasty (E-ESG), have shown effectiveness in weight loss and could offer a safer, more accessible alternative to surgery, in particular if associated to a lifestyle modifications program. Efficacy and safety of Bariatric endoscopy has been stressed within the recently published "Guideline of the Italian Society of Surgery of Obesity and Metabolic Diseases on Bariatric Endoscopy in the treatment of obesity and associated complications" that suggest the use of bariatric endoscopy in patients with class I obesity and in patients with class II obesity regardless of the presence of comorbidities, for the treatment of obesity.

This study aims to assess the feasibility and safety of the E-ESG procedure in treating obesity in women after curative treatment for endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometrial cancer scheduled for hysterectomy with a curative intent
* Age 21-75
* BMI ≥ 30
* Willingness to undergo E-ESG and lifestyle modifications program
* Willingness to comply with the substantial lifelong dietary restrictions required by the procedure
* Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, and completing diet counseling
* Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow- up visits
* Ability to give informed consent

Exclusion Criteria:

* History of foregut or gastrointestinal (GI) surgery (except uncomplicated cholecystectomy or appendectomy)
* Prior gastrointestinal surgery with sequelae, i.e., obstruction, and/or adhesive peritonitis or known abdominal adhesions
* Prior open or laparoscopic bariatric surgery
* Prior surgery of any kind on the esophagus, stomach, or any type of hiatal hernia surgery
* Any inflammatory disease of the gastrointestinal tract including severe (LA Grade C or D) esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease
* Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresia or stenoses
* Gastrointestinal stromal tumors, history of premalignant gastric lesions (advanced atrophic gastritis), history of familial and non-familial adenomatous syndromes
* A gastric mass or gastric polyps > 1 cm in size
* A hiatal hernia > 4 cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms
* A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope
* Achalasia or any other severe esophageal motility disorder
* Severe coagulopathy
* Subjects with any serious health condition unrelated to their weight that would increase the risk of endoscopy
* Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis, or intractable constipation
* Hepatic insufficiency or cirrhosis
* Use of an intragastric device prior to this study due to the increased thickness of the stomach wall preventing effective suturing
* Active psychological issues preventing participation in a life-style modification program as determined by a psychologist
* Patients unwilling to participate in an established medically supervised diet and behavior modification program, with routine medical follow-up
* Patients who are unable or unwilling to take prescribed proton pump inhibitor medication
* Patients receiving daily prescribed treatment with high dose aspirin (> 80 mg daily), anti-inflammatory agents, anticoagulants, or other gastric irritants
* Patients who are pregnant or breast-feeding
* Subjects with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs
* Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications
* Subjects who are taking corticosteroids, immunosuppressants, and narcotics
* Subjects who are taking diet pills
* Symptomatic congestive heart failure, cardiac arrhythmia, or unstable coronary artery disease
* Pre-existing respiratory disease such as moderate or severe chronic obstructive pulmonary disease (COPD) requiring steroids, pneumonia, or cancer
* Diagnosis of autoimmune connective tissue disorder (e.g., lupus, erythematosus, scleroderma) or immunocompromised
* Specific diagnosed genetic disorder such as Prader Willi syndrome
* Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating
* Known history of endocrine disorders affecting weight such as uncontrolled hypothyroidism

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with endometrial cancer scheduled for hysterectomy with a curative intent, with BMI ≥ 30 and Willingness to undergo E-ESG and lifestyle modifications program
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the feasibility of E-ESG procedure in obese patients with endometrial cancer. | up to 4 years
  Absolute and relative frequency of patients with technical success of E-ESG procedure, reported with relative 95% Confidence Interval

SECONDARY OUTCOMES:
Evaluation of patients who refused E-ESG procedure | up to 4 years
  Evaluation of the number and percentage of women with endometrial cancer and obese who refused E-ESG procedure
Evaluation of patients who refused E-ESG procedure | up to 4 years
  Description with absolute and relative frequencies of baseline characteristics of women with endometrial cancer and obese who refused E-ESG procedure
Evaluation of E-ESG safety in obese endometrial cancer patients. | up to 4 years
  Absolute and relative frequencies of adverse events
To evaluate efficacy of E-ESG effects on obesity-associated comorbidities. | up to 4 years
  Evaluation of % Excess weight loss (EWL) with the formula (Weight loss)/ (Excess weight at T0) x 100 and %TBWL(total body weight loss) with the formula (weight loss) / (weight at T0) x 100 in enrolled patients at 1 year
Evaluation of percentage of patients that reach a mean excess weight loss (EWL) of more than 25% and total body weight loss (TBWL) of more than 5% maintained at 1 year (52 weeks) in E-ESG and lifestyle modifications group | up to 4 years
  Absolute and relative frequencies of patients that reach a mean excess weight loss (EWL) of more than 25% and a total body weight loss (TBWL) of more than 5% maintained at 1 year (52 weeks)
To evaluate the change of metabolic serum biomarkers in E-ESG patients | up to 4 years
  Mean or median difference between baseline values of metabolic serum biomarkers and 52 weeks (T1), and 156 weeks (T2)
To evaluate the change of gut microbiota | up to 4 years
  Microbial levels will be described as mean or median, reporting differences in levels ad different time points
To evaluate Overall Survival in E-ESG | up to 4 years
  Overall survival will be defined as time between E-ESG and death from any cause or end of follow up, whichever cames first. Data will be described as median survival and interquartile range (IQR) calculated with Kaplan-Meyer method
To evaluate Disease Free Survival n E-ESG | up to 4 years
  Overall survival will be defined as time between E-ESG and disease progression or death from any cause or end of follow up, whichever cames first. Data will be described as median survival and interquartile range (IQR) calculated with Kaplan-Meyer method
To evaluate Recurrence rate in E-ESG | up to 4 years
  Disease recurrence rate at the end of follow up will be reported as absolute and relative frequency

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro di Riferimento Oncologico (CRO) - IRCCS Aviano, Aviano, Pordenone
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma, Roma